CLINICAL TRIAL: NCT03871335
Title: Work-related Musculoskeletal Disorders Among Female Workers in a Hazelnut Factory: Prevalence, Working Posture and Relating Factors
Brief Title: Work-related Musculoskeletal System Disorders Among Female Workers in Hazelnut Factory
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Collaborators: Giresun University (Other); Hacettepe University (Other)
Responsible Party: Principal Investigator, Sevim ACARÖZ CANDAN, Head of Department of Physiotherapy and Rehabilitation, PhD, Ordu University
Other Study IDs: OrduU4
Record Dates: First submitted 2019-02-11; First posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Musculoskeletal Strain; Pain; Occupational Problems; Work-related Injury
Keywords: work-related musculoskeletal disorders; hazelnut factory; low back pain; neck pain
MeSH Terms: conditions — Pain; Low Back Pain; Neck Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Investigation of the work-related musculoskeletal disorders — Structured questionnaires will be used to determine the prevalence of the work-related musculoskeletal disorders and work-related factor. Photogrammetric method will be used to evaluate working posture.

SUMMARY:
The aim of this study is to determine the prevalence of work-related musculoskeletal disorders in female workers in hazelnut factory. The secondary aim is to investigate the relationship between the musculoskeletal disorders severity and working posture, work related factor, psychosocial factor.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years,
* had at least 12 months of continuous working experience in hazelnut selection.

Exclusion Criteria:

* having pregnancy,
* working in a standing position or having a burden job,
* having joint disease, gout, diabetes, and trauma during the last one year

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of this study involved the female workers of a hazelnut factory.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2018-06-10 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Nordic Musculoskeletal Questionnaire (NMQ) | 10 minutes
  NMQ will be used to determine the self-reported musculoskeletal symptoms in the different body part (neck, shoulder, elbow, wrist, upper back, lower back, hip, knee, ankle) in which suffered from aches, pain, or discomfort during the last 12 months. The states of the obtained sick leave from work, obstructing of work, taken medication and seen a doctor or physiotherapist etc. during the past 12 months regarding the work-related MSD will be questioned. The participants can be responded by "yes" or "no".

SECONDARY OUTCOMES:
Dutch Musculoskeletal Questionnaire short version (DMQ-s) | 10 minutes
  DMQ-s was used to evaluate the perceived workload, work-related risk factors, and general health status. DMQ-s involves four sections (general question, health, perceived workload, ergonomic environment). The score of the three sections except the general questions section will be summed. Higher scores means risky situation for work-related musculoskeletal disorders.
Assessment of the working posture | 2 minutes
  The working posture will be assessed using the photogrammetry method which is a reliable and valid tool for postural angles analysis. The photographs were taken the lateral aspect of the workers using a digital, professional camera (Canon 4000D, Japan) from a 150cm distance, at the height of the acromion in working position. Cranio-vertebral angle (CVA), thoracic kyphosis and lumbar lordosis angles were measured on the photograph using the ImageJ program. The results will be recorded as degree.
Rapid Upper Extremity Assessment | 5 minutes
  Rapid Upper Limb Assessment (RULA) is a tool to evaluate upper extremity MSD risk factors. The RULA ergonomic assessment tool considers biomechanical and postural load requirements of job tasks/demands on the neck, trunk and upper extremities. A single page worksheet is used to evaluate required body posture, force, and repetition. Based on the evaluations, scores are entered for each body region in section A for the arm and wrist, and section B for the neck and trunk. After the data for each region is collected and scored, tables on the form are then used to compile the risk factor variables, generating a single score that represents the level of MSD risk. The score means 1-2 negligible risk no change requirement, 3-4 low risk change may be needed requirement, 5-6 medium risk further investigation change soon, 6+ very high risk implement change now
Short Form-12 Health Survey (SF-12 Health Survey) | 5 minutes
  SF-12 Health Survey is a multidimensional generic measure of health-related quality of life. SF-12 Health Survey includes two subdomains as physical and mental. SF-12 Health Survey has a scoring algorithm. The higher scores defines good quality of life.
Pain Severity | 5 minutes
  Pain severity will be scored between 0 and 10. The pain of nine different body part (neck, shoulder, elbow, wrist, upper back, lower back, hip, knee, ankle) will be examined by the subject's perception.

CONTACTS AND LOCATIONS:
Overall Officials: Sevim ACARÖZ CANDAN, Principal Investigator — Bayan
Locations (1):
- Sevim ACARÖZ CANDAN, Ordu, Altinordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No